CLINICAL TRIAL: NCT05627440
Title: A SkeleTal Muscle Recovery Intervention With Dietary Protein in Heart Failure
Acronym: ASTRID-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003095; 1R01HL167113-01 (NIH)
Record Dates: First submitted 2022-11-17; First posted 2022-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Muscle Atrophy
MeSH Terms: conditions — Heart Failure; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental arm (Experimental): 30 g/day protein supplementation (1 Ensure Max Protein® bottle)
  Interventions: Dietary Supplement: Ensure Max Protein
- Sham comparator arm (Active Comparator): 9 g/day protein supplementation (1 Ensure Original® bottle)
  Interventions: Dietary Supplement: Ensure Original
- No intervention arm (No Intervention): 0 g/day protein supplementation (no Ensure bottles)

INTERVENTIONS:
Dietary Supplement: Ensure Max Protein — Ensure Max Protein, 1 bottle daily (330 mL), 30 grams protein
  Arms: Experimental arm
Dietary Supplement: Ensure Original — Ensure Original, 1 bottle daily (237 mL), 9 grams protein
  Arms: Sham comparator arm

SUMMARY:
Severe skeletal wasting and catabolic weight loss are highly common among patients with heart failure with reduced ejection fraction (HFrEF). This prospective randomized controlled trial will compare changes in the muscle mass in the arms and the legs (appendicular lean mass) in patients with HFrEF randomized between 3 groups of no, low- or high-dose protein supplementation. The dietary protein supplementation will be Ensure(R) products manufactured by Abbott Nutrition. The Investigators hypothesize that skeletal muscle wasting in HFrEF is promoted by neurohumoral activation of catabolic metabolism (such as GDF-15 and ActRII pathways) and can be at least partially reversed by increased dietary protein intake. It is anticipated that this study will determine whether dietary protein supplementation helps to prevent muscle wasting and will advance understanding of the GDF-15 and ActRII muscle wasting pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Left ventricular ejection fraction (LVEF) ≤40%, New York Heart Association (NHYA) class II to IV symptoms or N-terminal pro B-natriuretic peptide (NT-proBNP) >300 pg/mL
2. Age 18 years to 100 years, inclusive
3. Receiving guideline-directed medical therapy (GDMT), unless contraindicated or not tolerated
4. Any of the following markers of severe HF within prior 12 months: i) Inotropic therapy; ii) 1 or more HF hospitalizations; iii) LVEF ≤25%; iv) Peak oxygen consumption (VO2) <50% predicted or ≤16 mL/kg/min; v) 6-minute walk distance <300 meters; vi) Unintentional weight loss >5% of bodyweight over the past year; vii) Moderate or severe muscle wasting on physical examination; viii) NT-proBNP ≥900 pg/mL

Exclusion Criteria:

1. Pregnancy, planning to become pregnant, or women of reproductive potential unwilling to complete pre-DXA urine pregnancy test before first DXA or randomization
2. History of left ventricular assist device (LVAD), heart transplantation, or estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2
3. An identified clinical disorder associated with skeletal muscle weakness/wasting (e.g., muscular dystrophy, mitochondrial disorder, active cancer, modified Rankin score greater or equal to 4 post-stroke)
4. Milk allergy, protein allergy, lactose intolerance, and galactosemia
5. Weight ≥350 pounds and/or BMI ≥40 kg/m2
6. Initiation of obesity-dosed GLP-1 or GIP/GLP-1 agonist within 3 months prior to screening, or clinical intention to begin such an anti-obesity medication within the next 6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Appendicular Lean Mass (ALM) | 6 month study visit
  ALM as measured by dual X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Appendicular Lean Mass (ALM) | 3 month study visit
  ALM as measured by dual X-ray absorptiometry (DXA)
Protein intake | 6 month study visit
  Dietary protein intake in g/kg/day, averaged over 3 days, which is calculated by entering recorded dietary intake from facilitate food record into the Food Processor® software
Protein intake | 3 month study visit
  Dietary protein intake in g/kg/day, averaged over 3 days, which is calculated by entering recorded dietary intake from facilitated food record into the Food Processor® software
Handgrip strength | 6 month study visit
  Strength in dominant hand assessed with 3 attempts using a hydraulic hand dynamometer in the dominant hand (Baseline® Evaluation Instruments Fabrication Enterprises Inc., Irvington NY) and the mean calculated
Handgrip strength | 3 month study visit
  Strength in dominant hand assessed with 3 attempts using a hydraulic hand dynamometer in the dominant hand (Baseline® Evaluation Instruments Fabrication Enterprises Inc., Irvington NY) and the mean calculated
6-minute walk test (6MWT) | 6 month study visit
  6-minute walk test measured over 100-foot laps, with 0 feet assigned if no independent ambulation is possible
6-minute walk test (6MWT) | 3 month study visit
  6-minute walk test measured over 100-foot laps, with 0 feet assigned if no independent ambulation is possible
Short physical performance battery (SPPB) | 6 months
  SPPB assesses balance, gait, strength, and endurance, by recording the ability to stand for up to 10 seconds with feet in the side-by-side, semi-tandem, and tandem positions; time to complete a 4-meter walk; and time to rise from a chair and return to the seated position 5 times
Short physical performance battery (SPPB) | 3 months
  SPPB assesses balance, gait, strength, and endurance, by recording the ability to stand for up to 10 seconds with feet in the side-by-side, semi-tandem, and tandem positions; time to complete a 4-meter walk; and time to rise from a chair and return to the seated position 5 times

OTHER OUTCOMES:
Fat free mass (FFM) | 6 months
  FFM as measured by dual X-ray absorptiometry (DXA)
Fat free mass (FFM) | 3 months
  FFM as measured by dual X-ray absorptiometry (DXA)
Fat mass (FM) | 6 months
  FM as measured by dual X-ray absorptiometry (DXA)
Fat mass (FM) | 3 months
  FM as measured by dual X-ray absorptiometry (DXA)
Weight | 6 months
  Bodyweight
Weight | 3 months
  Bodyweight
Simplified Nutritional Appetite Questionnaire (SNAQ) | 6 months
  Malnutrition risk assessment tool
Simplified Nutritional Appetite Questionnaire (SNAQ) | 3 months
  Malnutrition risk assessment tool
Mini-Nutritional Assessment-Short Form (MNA-SF) | 6 months
  Malnutrition risk assessment tool
Mini-Nutritional Assessment-Short Form (MNA-SF) | 3 months
  Malnutrition risk assessment tool
Subjective Global Assessment (SGA) | 6 months
  Semi-quantified assessment of cachexia per physical examination
Subjective Global Assessment (SGA) | 3 months
  Semi-quantified assessment of cachexia per physical examination
Growth Differentiation Factor (GDF)-15 | 3 months
  Inflammatory and growth regulation cytokine blood concentration
Growth Differentiation Factor (GDF)-15 | 6 months
  Inflammatory and growth regulation cytokine blood concentration
Activin A and Follistatin-related gene (FSTL)-3 | 3 months
  Muscle growth regulation pathway blood concentrations
Activin A and Follistatin-related gene (FSTL)-3 | 6 months
  Muscle growth regulation pathway blood concentrations

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plans will be reviewed by the Tufts Health Sciences IRB and no identifiable participant data will be shared outside Tufts Medical Center. A data use agreement (DUA) will be completed between the PI and collaborating sites.
Time Frame: After primary and secondary analyses have been completed and the major findings for each Aim accepted for publication.
Access Criteria: Due to the small sample size and single center location of the subjects, there remains a potential for deductive disclosure of subjects with unique clinical characteristics. Thus, the DUA will include language requiring: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.